CLINICAL TRIAL: NCT06910813
Title: An Open-label, Multi-center, Phase I/II Study to Assess Safety, Tolerability and Efficacy of DFT383 in Pediatric Participants With Nephropathic Cystinosis, Followed by a Long-term Extension Phase
Brief Title: DFT383 in Pediatric Participants With Nephropathic Cystinosis
Acronym: CYStem
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDFT383A12101
Record Dates: First submitted 2025-03-17; First posted 2025-04-04 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Nephropathic Cystinosis
Keywords: Cystinosis; Nephropathic cystinosis; Lysosomal storage disorder; CTNS gene; DFT383; Cellular gene therapy; Cysteamine; Renal Fanconi syndrome
MeSH Terms: conditions — Cystinosis; Lysosomal Storage Diseases; Fanconi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (DFT383) (Experimental): Treatment with DFT383
  Interventions: Genetic: DFT383
- Cohort 0 (SoC) (No Intervention): No study treatment, will continue with standard of care (cysteamine).

INTERVENTIONS:
Genetic: DFT383 — DFT383 is an autologous hematopoietic stem cell (HSC) gene therapy.
  Arms: Cohort 1 (DFT383)

SUMMARY:
An open-label, multi-center, phase I/II study to assess the safety, tolerability and efficacy of DFT383 in pediatric participants with nephropathic cystinosis, followed by a long-term extension phase.

The purpose of this clinical study is to assess safety, tolerability, and efficacy of DFT383 in participants aged 2 to 5 years with nephropathic cystinosis. The study consists of a Core Phase and a long-term Extension Phase. DFT383 is a cellular gene therapy.

This study includes an active arm (Cohort 1) of participants treated with study treatment DFT383 and a concurrent reference arm (Cohort 0). Participants in Cohort 0 will not receive study treatment and will only participate in the Core Phase of the study. The study is not randomized and Cohort 0 aims to collect prospective and concurrent data in this rare disease.

DETAILED DESCRIPTION:
This study is an open-label, multi-center, phase I/II study to assess the safety, tolerability, and efficacy of DFT383 in participants aged 2 to 5 years with nephropathic cystinosis, followed by a long-term extension phase.

The study includes two Treatment Groups (Cohort 1 and Cohort 0) and consists of a Core Phase and a long-term Extension Phase.

Participants in Cohort 1 will receive DFT383 and participate in both the Core and Extension Phase. Participants in Cohort 0 will not receive study treatment and will participate in the Core Phase only.

The two cohorts will be run in parallel. Investigational sites may participate in one or both cohorts.

Cohort 1 Approximately 15 participants will receive treatment with DFT383 in 3 (sub) cohorts (1A, 1B and 1C) dosed in a staggered approach. The total study duration for a participant in Cohort 1 will be up to 32 months in the core phase and up to 13 years for the long-term extension phase.

Cohort 0 Approximately 15 participants meeting similar inclusion/exclusion criteria and receiving SoC will be enrolled. The Schedule of Activities will be reduced for this Cohort. This cohort 0 is not a direct control but will provide essential context for interpreting the results observed in the participants receiving DFT383. The total study duration for a participant in Cohort 0 will be up to 24 months.

ELIGIBILITY:
Key Inclusion Criteria:

Participants eligible for inclusion in this study must meet all the following criteria:

1. Informed consent in writing from parent(s) or legal guardian(s) must be provided
2. 2 to 5 years of age (including 5 years and 364 days old) at Screening
3. Weight-for-stature is ≥ the third percentile, and is ≥ 10 kg
4. Oral cysteamine therapy for at least 6 months
5. Historic clinical diagnosis of nephropathic cystinosis
6. Laboratory evidence of of renal fanconi syndrome (RFS)
7. Relatively preserved kidney function (eGFR ≥ 60mL/min/1.73m2)
8. Received all age-appropriate vaccinations

Key exclusion Criteria for Cohort 1 and 0

1. A history of kidney transplantation
2. A prior or planned bone marrow or stem cell transplantation or prior treatment with gene therapy
3. History of malignancy
4. A severe or uncontrolled medical disorder
5. Major surgery within 90 days

Additional Key exclusion criteria for Cohort 1 - The following exclusion criterion applies to Cohort 1 only as it is related to DFT383 treatment:

1. Indomethacin within 2 weeks prior to Screening

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2031-03-14 (Estimated); Study Completion 2044-03-14 (Estimated)

PRIMARY OUTCOMES:
Core Phase - Incidence of adverse events (Cohort 1) | Up to 32 months
  Number and proportion of participants with adverse events (AEs) and serious adverse events (SAEs)
Core Phase - Number of participants with hematological reconstitution (Cohort 1) | 42 days post DFT infusion
  Hematological reconstitution by Day 42 post-DFT383 infusion
Core Phase - Proportion of participants with reversal of renal Fanconi syndrome (RFS) | Up to 32 months
  Proportion of participants with reversal of renal Fanconi syndrome (RFS)

SECONDARY OUTCOMES:
Core Phase - Number of participants independent from cysteamine | up to 24 months
  Independence from oral and ophthalmic cysteamine
Core Phase - Health-related quality of life (HRQOL) | Up to 32 months
  Health-related quality of life (HRQOL) as measured by QUALIFY (cystinosis-specific PRO)- Currently under development
Core Phase - Time from infusion to reversal of RFS (Cohort 1) | Up to 24 months
  Time from infusion to reversal of renal Fanconi syndrome (RFS)
Core Phase - Time from screening to reversal of RFS (Cohort 0) | Up to 24 months
  Time from screening to reversal of renal Fanconi syndrome (RFS)
Core Phase - Duration of reversal of RFS | Up to 24 months
  Duration of reversal of renal Fanconi syndrome (RFS)
Core Phase - Change from baseline on urine protein to creatinine ratio (UPr/CR) | Up to 27 months
  Change from baseline on urine protein to creatinine ratio (UPr/CR)
Core Phase - Change from baseline on urine amino acids | Up to 27 months
  Change from baseline on urine amino acids
Core Phase - Change from baseline on urinary glucose to creatinine ratio | Up to 27 months
  Change from baseline on urinary glucose to creatinine ratio
Core Phase - Change from baseline on tubular maximum reabsorption of Phosphate/Glomerular Filtration Rate ratio (TmP/GFR) | Up to 27 months
  Change from baseline on tubular maximum reabsorption of Phosphate/Glomerular Filtration Rate ratio
Core Phase - Change from baseline on urine retinol-binding protein/creatinine ratio (RBP/Cr) | Up to 27 months
  Change from baseline on urine retinol-binding protein/creatinine ratio
Core Phase - Number of participants with improvement of proximal tubular function | Up to 27 months
  Improvement of proximal tubular function as defined by 2-fold change from Baseline of at least 4 out of 5 RFS parameters (urine protein to creatinine ratio, urine amino acids, urinary glucose to creatinine ratio, tubular maximum reabsorption of Phosphate/Glomerular Filtration Rate, urine retinol-binding protein/creatinine ratio). Improvement will also be considered if the change from Baseline is less than 2-fold but the value falls within the definition for normalization.
Core Phase - Corneal cystine crystal content | Up to 27 months
  Corneal crystal content by anterior segment optical coherence tomography (AS-OCT)
Core Phase - Number of participants with clinically significant changes in vital signs, physical examinations, laboratories, and ECG (Cohort 1) | Up to 27 months
  Vital signs, physical examinations, laboratories (eg., chemistry, hematology, liver function tests), and ECG
Core Phase - Number of participants with presence/emergence of replication-competent lentivirus (Cohort 1) | Up to 27 months
  Number of participants with presence/emergence of replication-competent lentivirus
Core Phase - Number of participants with malignancy (Cohort 1) | Up to 27 months
  Number of participants with malignancy
Core Phase - Time to hematological reconstitution (Cohort 1) | Up to 24 months
  Time to hematological reconstitution
Core Phase - Time to platelet engraftment (Cohort 1) | Up to 24 months
  Time to platelet engraftment
Core Phase - Incidence of Adverse Events (Cohort 0) | up to 24 months
  Number and proportion of participants with adverse events (AEs) and serious adverse events (SAEs)
Extension Phase Primary Objective - Incidence of Adverse events (Cohort 1) | Up to 15 years and 8 months
  Number and proportion of participants with adverse events (AEs) and serious adverse events (SAEs)
Extension Phase - Number of participants with malignancy (Cohort 1) | Up to 15 years and 3 months
  Number of participants with malignancy
Extension Phase - Number of participants with presence/emergence of replication-competent lentivirus (Cohort 1) | Up to 15 years and 3 months
  Number of participants with presence/emergence of replication-competent lentivirus
Extension Phase - Number of participants with clinically significant changes in vital signs, physical examinations, laboratories, and ECG (Cohort 1) | Up to 15 years and 3 months
  Vital signs, physical examinations, laboratories (eg., chemistry, hematology, liver function tests), and ECG
Extension Phase - Change from baseline on urine protein to creatinine ratio (UPr/CR) (Cohort 1) | Up to 15 years and 3 months
  Change from baseline on urine protein to creatinine ratio (UPr/CR)
Extension Phase - Change from baseline on urine amino acids (Cohort 1) | Up to 15 years and 3 months
  Change from baseline on urine amino acids
Extension Phase - Change from baseline on urinary glucose to creatinine ratio (Cohort 1) | Up to 15 years and 3 months
  Change from baseline on urinary glucose to creatinine ratio
Extension Phase - Change from baseline on tubular maximum reabsorption of Phosphate/Glomerular Filtration Rate ratio (TmP/GFR) (Cohort 1) | Up to 15 years and 3 months
  Change from baseline on tubular maximum reabsorption of Phosphate/Glomerular Filtration Rate ratio
Extension Phase - Change from baseline on urine retinol-binding protein/creatinine ratio (RBP/Cr) (Cohort 1) | Up to 15 years and 3 months
  Change from baseline on urine retinol-binding protein/creatinine ratio
Extension Phase - Duration of reversal of RFS (Cohort 1) | Up to 15 years
  Duration of reversal of renal Fanconi syndrome (RFS)
Extension Phase - Number of participants with kidney failure (Cohort 1) | Up to 15 years
  Number of participants with kidney failure
Extension Phase - Number of participants independent from cysteamine (Cohort 1) | Up to 15 years
  Independence from oral and ophthalmic cysteamine
Extension Phase - Corneal cystine crystal content (Cohort 1) | Up to 15 years and 3 months
  Corneal crystal content by anterior segment optical coherence tomography (AS-OCT)
Extension Phase - Health-related quality of life (HRQOL) (Cohort 1) | Up to 15 years and 8 months
  Health-related quality of life (HRQOL) as measured by QUALIFY (cystinosis-specific PRO)- Currently under development

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of California at San Diego - Rady Children's Hospital, San Diego, California
  - Stanford University - Stanford Children's Health, Stanford, California
  - Emory University School of Medicine - Children's Healthcare of Atlanta (recuiting Cohort 0), Atlanta, Georgia
  - Baylor College of Medicine - Texas Children's Hospital (recuiting Cohort 0), Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes